CLINICAL TRIAL: NCT02883036
Title: Changes of Mitochondrial Biogenesis and Metabolic Characteristics About Tigecycline to Treat Chronic Myeloid Leukemia in Vitro
Brief Title: Vitro Study of Tigecycline to Treat Chronic Myeloid Leukemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Xiaoli Liu, professor, Nanfang Hospital, Southern Medical University
Other Study IDs: VSTICML-01
Record Dates: First submitted 2016-08-19; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Myeloid Leukemia
Keywords: tigecycline; treatment; mitochondrial biogenesis; metabolic characteristics
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — mononuclear cells of bone marrow and/or peripheral blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with chronic myeloid leukemia: 100 adult patients(age>18 years),with chronic myeloid leukemia defined by the World Health Organization(WHO) criteria
  Interventions: Other: blood sampling
- Healthy volunteers: Healthy volunteers
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — sampling after diagnosis and the mononuclear cells will be given tigecycline stimulation in vitro
  Groups: Patients with chronic myeloid leukemia
Other: blood sampling — sampling after register and the mononuclear cells will be given tigecycline stimulation in vitro
  Groups: Healthy volunteers

SUMMARY:
Chronic myeloid leukemia (CML) is a myeloproliferative neoplasm companies with the BCR-ABL fusion gene encoded by the Philadelphia (Ph) chromosome. The BCR-ABL fusion protein(the formation of the chimeric gene BCR/ABL on chromosome 22 and a reciprocal ABL/BCR on chromosome 9,it has no expanded name) plays key role on CML leukemogenesis by activating its downstream signaling pathway of survival and proliferation. Imatinib, a targeted competitive inhibitor of a BCR-ABL tyrosine kinase, changed the clinical treatment and prognosis of CML. As its optimized generation, other tyrosine kinase inhibitors (TKIs), dasatinib and nilotinib have more potent anti-leukemic activity and less side-effect. However, acquired resistance to TKIs is one of the main obstacles to effective CML treatment and is involved in gene amplication of ABL tyrosine kinase point mutations. The outcomes of patients with these ABL tyrosine kinase point mutations have linked to worse prognosis and higher mortality generally. Metabolic adaptations are common in cancer cells, and cancer cells become more dependent on mitochondrial biogenesis. Tigecycline, as a broad-spectrum antibiotics, inhibits mitochondrial biogenesis as its an interesting "side-effect".In recent study,researchers indicated that tigecycline can eradicate cancer stem cells by targeting mitochondrial.Here, the investigators test tigecycline's anti-leukemic activity to chronic myeloid leukemia in vitro.

DETAILED DESCRIPTION:
In this study, the investigators collected bone marrow(BM) or/and peripheral blood(PB) mononuclear cells from patients with chronic myeloid leukemia.Patients could be in different stages of chronic myeloid leukemia pre-treatment.Additionally, the investigators also selected some healthy volunteers as comparison.Firstly, the investigators analyzed mitochondrial biogenesis and basal metabolic characteristic of mononuclear cells from patients and healthy volunteers.Secondly, the investigators tested the cell viability and apoptosis after tigecycline treatment.Thirdly,the investigators detected the changes of cell mitochondrial biogenesis and metabolic characteristic in the same study sample after tigecycline stimulation. Finally,the investigators analyzed the correlation between sensitivities of mononuclear cells to tigecycline and patients' clinical parameters and survival outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Philadelphia chromosome positive and/or BCR-ABL positive CML confirmed by cytogenetic and/or molecular analysis;
* Age >18 years.
* Eligibility of patients receiving any medications or substances known to affect or determined following review of their case by the Principal Investigator

Exclusion Criteria:

* Patients may not receive any other antibiotics.
* Patients may not have received prior treatment with TKIs or hydroxyurea.
* Major cognitive deficits or psychiatric problems hampering a self-reported evaluation.
* No prior malignancies or any other cancer from which patient has been disease free for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 adults patients with chronic myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
mitochondrial biogenesis and metabolic characteristics of Bone Marrow(BM)/ Peripheral Blood(PB) mononuclear cells | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
mitochondrial biogenesis and metabolic characteristics of BM/PB mononuclear cells after tigecycline stimulation | After Hour 24 and 48 tigecycline stimulation
cell viability and apoptosis of BM/PB mononuclear cells after tigecycline stimulation | After Hour 24 and 48 tigecycline stimulation
Patients' clinical characteristics and survival outcomes | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of hematology,Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lamb R, Ozsvari B, Lisanti CL, Tanowitz HB, Howell A, Martinez-Outschoorn UE, Sotgia F, Lisanti MP. Antibiotics that target mitochondria effectively eradicate cancer stem cells, across multiple tumor types: treating cancer like an infectious disease. Oncotarget. 2015 Mar 10;6(7):4569-84. doi: 10.18632/oncotarget.3174. PMID 25625193
- [Background] Skrtic M, Sriskanthadevan S, Jhas B, Gebbia M, Wang X, Wang Z, Hurren R, Jitkova Y, Gronda M, Maclean N, Lai CK, Eberhard Y, Bartoszko J, Spagnuolo P, Rutledge AC, Datti A, Ketela T, Moffat J, Robinson BH, Cameron JH, Wrana J, Eaves CJ, Minden MD, Wang JC, Dick JE, Humphries K, Nislow C, Giaever G, Schimmer AD. Inhibition of mitochondrial translation as a therapeutic strategy for human acute myeloid leukemia. Cancer Cell. 2011 Nov 15;20(5):674-88. doi: 10.1016/j.ccr.2011.10.015. PMID 22094260